CLINICAL TRIAL: NCT04366323
Title: Phase I / II Clinical Trial, Multicenter, Randomized and Controlled, to Assess the Safety and Efficacy of Intravenous Administration of Allogeneic Adult Mesenchymal Stem Cells of Expanded Adipose Tissue in Patients With Severe Pneumonia Due to COVID-19
Brief Title: Clinical Trial to Assess the Safety and Efficacy of Intravenous Administration of Allogeneic Adult Mesenchymal Stem Cells of Expanded Adipose Tissue in Patients With Severe Pneumonia Due to COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdiQure/COVID-19
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Sars-CoV2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: ALLOGENEIC AND EXPANDED ADIPOSE TISSUE-DERIVED MESENCHYMAL STEM CELLS
- Control (No Intervention)

INTERVENTIONS:
Drug: ALLOGENEIC AND EXPANDED ADIPOSE TISSUE-DERIVED MESENCHYMAL STEM CELLS — Two doses of 80 million adipose-tissue derived mesenchymal stem cells
  Arms: Experimental

SUMMARY:
Phase I/II clinical trial to evaluate the safety and efficacy of Allogenic Adipose Tissue-Derived Mesenchymal Stem Cells Expanded in patients with severe COVID-19 pneumonia

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Clinical diagnosis of Pneumonia, severe or critical, caused by COVID-19 infection
3. Life expectancy > 48 hours.
4. Commitment to use a contraceptive method of proven efficacy in both men and women during the duration of the clinical trial.

Exclusion Criteria:

1. Coinfection with other viruses or bacteria (HIV, tuberculosis, influenza virus, adenovirus or other respiratory infections, active infection by HBV or C).
2. History of multiple allergies, including allergy to Penicillin or other Blactams.
3. Pregnant and lactating women.
4. Patients with malignant tumors or hemopathies or any state of immunosuppression considered as severe.
5. Patients with autoimmune diseases.
6. Chronic heart failure with ejection fraction less than 30%.
7. Any other condition for which, in the opinion of the main investigator, the subject is considered not to be in compliance with the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Safety of the administration of allogeneic mesenchymal stem cells derived from adipose tissue assessed by Adverse Event Rate | 12 months
Efficacy of the administration of allogeneic mesenchymal stem cells derived from adipose tissue assessed by Survival Rate | 28 days

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Unversitario Virgen del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville

IPD SHARING:
Plan to Share IPD: No